CLINICAL TRIAL: NCT04168801
Title: Non-inferiority Comparative Clinical Trial Between Early Oral Refeeding Versus Usual Oral Refeeding in Mild Acute Pancreatitis Patients
Brief Title: Early Oral Refeeding in Mild Acute Pancreatitis
Acronym: EORVsUOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Regional de Alta Especialidad del Bajio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hraeb; EORvsUOR project (Registry Identifier: EORvsUOR project)
Record Dates: First submitted 2019-11-07; First posted 2019-11-19 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Pancreatitis
Keywords: Mild acute pancreatitis; Oral refeeding; Non inferiority clinical trial
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Intervention Model Description: Prior authorization from the ethics committee in health research. Patients with diagnosis of mild acute biliary pancreatitis, were divided into: Group A (early oral refeeding) and Group B (usual oral refeeding). Outcome measures were lipase pancreatic, systemic inflammatory response (concentrations of leukocytes) were used as marker for it, feasibility evaluated by abdominal pain recurrence, presence and recurrence of gastrointestinal symptoms and length of hospital stay.
Who Masked: Outcomes Assessor
Masking Description: Only the person who performed the statistical analysis did not know to which group each patient belonged
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early oral refeeding (Experimental): Once the patient had a score of 1-3 of the analogue numerical scale (ENA), he was interrogated about symptoms such as nausea or vomiting, if he did not have them, then receives diet indicated between 16 and 24 hours after admission.
  Interventions: Dietary Supplement: early oral refeeding
- Usual oral refeeding (Active Comparator): usual oral refeeding (UOR) Once the attending physician decided according to his clinical judgment to restart the oral feeding
  Interventions: Dietary Supplement: early oral refeeding

INTERVENTIONS:
Dietary Supplement: early oral refeeding — Once the patient had a score of 1-3 of the analogue numerical scale (ENA), he was interrogated about symptoms such as nausea or vomiting, receives diet indicated between 16 and 24 hours after admission.
  Other Names: Early Vs Usual oral refeeding

SUMMARY:
Background The aim of the study is to compare the onset of oral feeding in the first 24 hours after hospital admission and determine if this influences the recurrence of pain or alters the blood levels of pancreatic enzymes, compared to usual oral refeeding in patients with mild acute pancreatitis Methods This Non-Inferiority Randomized controlled trial was carried out between September 2018 and June 2019, prior authorization from the ethics committee in health research. Patients with diagnosis of mild acute biliary pancreatitis, were divided into: Group A (early oral refeeding) and Group B (usual oral refeeding). Outcome measures were lipase pancreatic, systemic inflammatory response (concentrations of leukocytes) were used as marker for it, feasibility evaluated by abdominal pain recurrence, presence and recurrence of gastrointestinal symptoms and length of hospital stay. The aim of the present study is to compare the onset of oral feeding in the first 24 hours after hospital admission and determine if this influences the recurrence of pain or alters the blood levels of pancreatic enzymes, compared to usual oral refeeding in patients with mild acute pancreatitis.

DETAILED DESCRIPTION:
BACKGROUND Acute pancreatitis (AP) is an inflammatory pancreatic process, presents different severity degrees [1]. Over the last two decades, there has been a paradigm shift in the management, from surgical to "step up" approach using percutaneous or endoscopic catheter drainage followed by minimally invasive necrosectomy [2]. As no curative therapy is currently available for AP, early treatment consists of supportive care which includes adequate fluid resuscitation, pain management and enteral nutrition [3]. Pancreatic rest by Nil Per Oral (NPO) strategy was considered necessary in AP till abdominal pain get resolved and the levels of pancreatic and inflammatory markers decrease [4]. This trend has changed, now it is clear that the early oral refeeding for PA mild does not only provide adequate caloric intake, it may also improve clinical outcomes. It has been hypothesized that the combination of disturbed intestinal motility, microbial overgrowth and increased permeability of the gut can lead to bacterial translocation, thus causing infection of pancreatic necrosis [5,6].

The oral refeeding (OR) may reduce translocation by stimulating intestinal motility, reducing bacterial overgrowth and thereby maintaining mucosal gut integrity [7,8]. Also decrease infection complications, organ failure and mortality as compared with routine total parenteral nutrition [9,10]. In patients with (predicted) mild pancreatitis, numerous studies concluded that a normal oral diet can be resumed once the pain is decreasing [11-13], However, it remains unclear what the optimal time to do it is. There is still no consensus about the definition of "early" refeeding.

The aim of the present study is to compare the onset of oral feeding in the first 24 hours after hospital admission and determine if this influences the recurrence of pain or alters the blood levels of pancreatic enzymes, compared to usual oral refeeding in patients with mild acute pancreatitis.

METHODS

Patients This Randomized controlled trial was carried out between September 2018 and June 2019, prior authorization from the ethics committee in health research.

A total number of 124 patients were randomized in this study. The sample size was calculated according to the formula published by Bouemn et all 2015 [14], in which a percentage of success was estimated with the standard treatment of 90% compared to the experimental management of 85%, with a margin of no less than 10%, with an alpha for a tail of 0.05%, and a beta of 20 %, with a percentage of estimated losses of approximately 10%, a total of 62 patients per group was obtained.

Definitions The diagnosis of AP was established when the patient presents two or more of the following three findings: typical abdominal pain, elevation of serum pancreatic enzymes (amylase and/or lipase) at more than three times the upper limit of the normal value, and imaging study (ultrasonography or computed tomography) suggestive of AP [15].

Severity Assessment Severity assessment of AP was done based on the revised Atlanta classification into mild, moderately severe and severe. Absence of organ failure or local or systemic complications was labelled as mild AP; of was defined using the modified Marshall scoring system [16]; and only the patients whose complete these severity criteria were randomized for the study.

Protocol Once the diagnosis of acute biliary pancreatitis was confirmed and the course was mild, corresponding informed consent signed.

Fluid therapy with crystalloid solution (Hartmann), initial bolus of 10 mL / kg and followed by infusion for 24 h of 1.5 mL / kg / h.

Pain management with opioid weak tramadol 50mg every 6 hours and paracetamol 1 gram every 8 hours with continuous evaluation of the analogue numerical scale to determine the need for extra doses

Type of Diet:

In both groups, their initial diet was the same so that this did not influence the results to be measured.

The soft diet consisted of one of 900 Kcal per day, with 86.7% carbohydrates (190 g), 13.3% protein (30 g) and 0% lipids (0 g); during 24 h.

When the diet was adequately tolerated and there was no evidence of clinical complications or deterioration, normal diet was indicated, and the follow-up continues.

Data Collection:

Laboratorial data, such as leukocytes, amylase and lipase were collected after inclusion in the study and after 24 and 48 h of oral refeeding. Clinical data records include age, gender, time from onset of pain baseline, Marshall score at admission and after start the oral feeding, gastrointestinal symptoms, abdominal pain, days until solid food intake, pain relapse, complications, length of hospital stay and readmissions.

Statistical analysis Date are presented as frequency and percentage, comparisons between groups were using the χ2 test for binary data or Fisher´s exact test. Continuous variables are presented as median and range interquartile range and were compared using the Mann-Whitney U-test or t student test if they meet normal criteria. p-Values of less than 0.05 were considered significant. Statistical analyses were performed with SPSS version 25.0.0. Analysis by intention to treat was used.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the surgery services with diagnosis of acute biliary pancreatitis
* Whit mild episode criteria and symptom onset time less than 24 hours

Exclusion Criteria:

* Patients with pancreatitis from another cause other than biliary
* Pregnant
* History of chronic pancreatitis
* Under 18 or over 75 years
* With moderately severe or severe acute biliary pancreatitis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-20 (Actual)

PRIMARY OUTCOMES:
abdominal pain recurrence | 72 hours
  Presence of abdominal pain after to oral refeeding

SECONDARY OUTCOMES:
systemic inflammatory response | 72 hours
  presence of systematic inflammatory response syndrome data, fever, leukocytosis

CONTACTS AND LOCATIONS:
Overall Officials: Edgard Lozada, Dr, Principal Investigator — Hospital Regional de Alta Especialidad
Locations (1):
- Hospital Regional de Alta Especilidad del bajio, León, Guanajuato, Mexico

IPD SHARING:
Plan to Share IPD: Yes
the database will be made available to corroborate results.
Supporting Information: Study Protocol, ICF
Time Frame: 1 year
Access Criteria: will be sent via e-mail as soon as requested

REFERENCES:
- [Background] Li JY, Yu T, Chen GC, Yuan YH, Zhong W, Zhao LN, Chen QK. Enteral nutrition within 48 hours of admission improves clinical outcomes of acute pancreatitis by reducing complications: a meta-analysis. PLoS One. 2013 Jun 6;8(6):e64926. doi: 10.1371/journal.pone.0064926. Print 2013. PMID 23762266
- [Background] Samanta J, Rana A, Dhaka N, Agarwala R, Gupta P, Sinha SK, Gupta V, Yadav TD, Kochhar R. Ascites in acute pancreatitis: not a silent bystander. Pancreatology. 2019 Jul;19(5):646-652. doi: 10.1016/j.pan.2019.06.004. Epub 2019 Jun 9. PMID 31301995
- [Background] van Dijk SM, Hallensleben NDL, van Santvoort HC, Fockens P, van Goor H, Bruno MJ, Besselink MG; Dutch Pancreatitis Study Group. Acute pancreatitis: recent advances through randomised trials. Gut. 2017 Nov;66(11):2024-2032. doi: 10.1136/gutjnl-2016-313595. Epub 2017 Aug 24. PMID 28838972
- [Background] Chebli JM, Gaburri PD, Chebli LA. Oral refeeding in mild acute pancreatitis: an old challenge. World J Gastrointest Pathophysiol. 2011 Dec 15;2(6):100-2. doi: 10.4291/wjgp.v2.i6.100. PMID 22180843
- [Background] Ammori BJ, Leeder PC, King RF, Barclay GR, Martin IG, Larvin M, McMahon MJ. Early increase in intestinal permeability in patients with severe acute pancreatitis: correlation with endotoxemia, organ failure, and mortality. J Gastrointest Surg. 1999 May-Jun;3(3):252-62. doi: 10.1016/s1091-255x(99)80067-5. PMID 10481118
- [Background] Fritz S, Hackert T, Hartwig W, Rossmanith F, Strobel O, Schneider L, Will-Schweiger K, Kommerell M, Buchler MW, Werner J. Bacterial translocation and infected pancreatic necrosis in acute necrotizing pancreatitis derives from small bowel rather than from colon. Am J Surg. 2010 Jul;200(1):111-7. doi: 10.1016/j.amjsurg.2009.08.019. PMID 20637344
- [Background] Marik PE. What is the best way to feed patients with pancreatitis? Curr Opin Crit Care. 2009 Apr;15(2):131-8. doi: 10.1097/MCC.0b013e328319910a. PMID 19300086
- [Background] McClave SA, Heyland DK. The physiologic response and associated clinical benefits from provision of early enteral nutrition. Nutr Clin Pract. 2009 Jun-Jul;24(3):305-15. doi: 10.1177/0884533609335176. PMID 19483060
- [Background] Yi F, Ge L, Zhao J, Lei Y, Zhou F, Chen Z, Zhu Y, Xia B. Meta-analysis: total parenteral nutrition versus total enteral nutrition in predicted severe acute pancreatitis. Intern Med. 2012;51(6):523-30. doi: 10.2169/internalmedicine.51.6685. Epub 2012 Mar 15. PMID 22449657
- [Background] Leppaniemi A, Tolonen M, Tarasconi A, Segovia-Lohse H, Gamberini E, Kirkpatrick AW, Ball CG, Parry N, Sartelli M, Wolbrink D, van Goor H, Baiocchi G, Ansaloni L, Biffl W, Coccolini F, Di Saverio S, Kluger Y, Moore E, Catena F. 2019 WSES guidelines for the management of severe acute pancreatitis. World J Emerg Surg. 2019 Jun 13;14:27. doi: 10.1186/s13017-019-0247-0. eCollection 2019. PMID 31210778
- [Background] Eckerwall GE, Tingstedt BB, Bergenzaun PE, Andersson RG. Immediate oral feeding in patients with mild acute pancreatitis is safe and may accelerate recovery--a randomized clinical study. Clin Nutr. 2007 Dec;26(6):758-63. doi: 10.1016/j.clnu.2007.04.007. Epub 2007 Aug 24. PMID 17719703
- [Background] Moraes JM, Felga GE, Chebli LA, Franco MB, Gomes CA, Gaburri PD, Zanini A, Chebli JM. A full solid diet as the initial meal in mild acute pancreatitis is safe and result in a shorter length of hospitalization: results from a prospective, randomized, controlled, double-blind clinical trial. J Clin Gastroenterol. 2010 Aug;44(7):517-22. doi: 10.1097/MCG.0b013e3181c986b3. PMID 20054282
- [Background] Teich N, Aghdassi A, Fischer J, Walz B, Caca K, Wallochny T, von Aretin A, von Boyen G, Gopel S, Ockenga J, Leodolter A, Ruddel J, Weber E, Mayerle J, Lerch MM, Mossner J, Schiefke I. Optimal timing of oral refeeding in mild acute pancreatitis: results of an open randomized multicenter trial. Pancreas. 2010 Oct;39(7):1088-92. doi: 10.1097/MPA.0b013e3181d3ce05. PMID 20357692
- [Background] Bouman AC, ten Cate-Hoek AJ, Ramaekers BL, Joore MA. Sample Size Estimation for Non-Inferiority Trials: Frequentist Approach versus Decision Theory Approach. PLoS One. 2015 Jun 15;10(6):e0130531. doi: 10.1371/journal.pone.0130531. eCollection 2015. PMID 26076354
- [Background] Banks PA, Bollen TL, Dervenis C, Gooszen HG, Johnson CD, Sarr MG, Tsiotos GG, Vege SS; Acute Pancreatitis Classification Working Group. Classification of acute pancreatitis--2012: revision of the Atlanta classification and definitions by international consensus. Gut. 2013 Jan;62(1):102-11. doi: 10.1136/gutjnl-2012-302779. Epub 2012 Oct 25. PMID 23100216
- [Background] Marshall JC, Cook DJ, Christou NV, Bernard GR, Sprung CL, Sibbald WJ. Multiple organ dysfunction score: a reliable descriptor of a complex clinical outcome. Crit Care Med. 1995 Oct;23(10):1638-52. doi: 10.1097/00003246-199510000-00007. PMID 7587228
- [Background] Working Group IAP/APA Acute Pancreatitis Guidelines. IAP/APA evidence-based guidelines for the management of acute pancreatitis. Pancreatology. 2013 Jul-Aug;13(4 Suppl 2):e1-15. doi: 10.1016/j.pan.2013.07.063. PMID 24054878
- [Background] Larino-Noia J, Lindkvist B, Iglesias-Garcia J, Seijo-Rios S, Iglesias-Canle J, Dominguez-Munoz JE. Early and/or immediately full caloric diet versus standard refeeding in mild acute pancreatitis: a randomized open-label trial. Pancreatology. 2014 May-Jun;14(3):167-73. doi: 10.1016/j.pan.2014.02.008. Epub 2014 Mar 14. PMID 24854611
- [Background] Meng WB, Li X, Li YM, Zhou WC, Zhu XL. Three initial diets for management of mild acute pancreatitis: a meta-analysis. World J Gastroenterol. 2011 Oct 7;17(37):4235-41. doi: 10.3748/wjg.v17.i37.4235. PMID 22072857
- [Background] Horibe M, Nishizawa T, Suzuki H, Minami K, Yahagi N, Iwasaki E, Kanai T. Timing of oral refeeding in acute pancreatitis: A systematic review and meta-analysis. United European Gastroenterol J. 2016 Dec;4(6):725-732. doi: 10.1177/2050640615612368. Epub 2015 Oct 13. PMID 28408989
- [Derived] Lozada-Hernandez EE, Barron-Gonzalez O, Vazquez-Romero S, Cano-Rosas M, Apolinar-Jimenez E. Non-inferiority comparative clinical trial between early oral REFEEDING and usual oral REFEEDING in predicted mild acute biliary pancreatitis. BMC Gastroenterol. 2020 Jul 16;20(1):228. doi: 10.1186/s12876-020-01363-3. PMID 32677891

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-09-05): https://cdn.clinicaltrials.gov/large-docs/01/NCT04168801/Prot_SAP_ICF_000.pdf